CLINICAL TRIAL: NCT00316134
Title: Evaluation of Multiple Biomarkers in Serum and Pleural Fluid to Estimate the Probability of Cancer in Patients Presenting With an Undiagnosed Pleural Effusion
Brief Title: Multiple Biomarkers in Undiagnosed Pleural Effusion
Status: Terminated | Type: Observational
Why Stopped: The study was terminated on completion of the Pilot Study phase.
Sponsor: Fujirebio Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FDI-02 Pleural Effusion Study
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Pleural Effusion; Pleural Effusion, Malignant
Keywords: Pleural Diseases; Pleural Effusion; Pleural Effusion, Malignant; Pleural Neoplasms; Neoplasms, Pleural
MeSH Terms: conditions — Pleural Effusion; Pleural Effusion, Malignant; Pleural Diseases; Pleural Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and pleural fluids
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pts scheduled to remove pleural fluid
  Interventions: Procedure: Procedure/Surgery

INTERVENTIONS:
Procedure: Procedure/Surgery — Diagnostic and/or therapeutic procedure to remove pleural fluid.

SUMMARY:
The purpose of this clinical trial is to evaluate the ability of various biomarkers measured in serum and/or pleural fluids to estimate the risk of finding cancer in patients with undiagnosed pleural effusions. An algorithm for prediction of the risk of finding cancer in the patient using an optimal combination of markers will be developed, and patients will be categorized as having a low, moderate, or high risk of finding cancer that might be used to more effectively triage patients.

DETAILED DESCRIPTION:
Approximately 1.6 million cases of pleural effusion are seen in the US per year, with ~210,000 of those cases due to underlying malignancy. Pleural fluids have traditionally been divided into two types: transudative and exudative. The most common causes of transudative pleural effusion are congestive heart failure and cirrhosis. Common causes of exudative pleural effusion include malignancy, pneumonia, pulmonary embolism and viral infection. One study found that 42% of all exudative effusions were due to malignancy, and another found that malignancy was the underlying cause of 24% of all effusions. Differential diagnosis of the various causes of effusions is complex and includes gross appearance of the pleural fluid (PF), differential cell count, cytology, glucose and LDH levels, and sometimes adenosine deaminase (ADA) levels. In addition, spiral CT scans, bronchoscopy, thoracoscopy, needle biopsy of the pleura, and video assisted thoracoscopy (VATS) are all utilized to determine the underlying cause of pleural fluid accumulation. These procedures are expensive and may be traumatic to patients. In approximately 20% of patients presenting with pleural fluid accumulation, no underlying cause will be established. Despite promising results published in peer-reviewed journals over the last two decades, serum biomarkers have not gained acceptance as a standard of care in the management of patients with lung cancer, mesothelioma, or pleural effusion. The purpose of this clinical trial is to evaluate the ability of various biomarkers measured in serum and/or pleural fluids to estimate the risk of finding cancer in patients with undiagnosed pleural effusions. An algorithm for prediction of the risk of finding cancer in the patient using an optimal combination of markers will be developed, and patients will be categorized as having a low, moderate, or high risk of finding cancer that might be used to more effectively triage patients. For example, a high risk of cancer may be used to justify more invasive or expensive procedures, such as spiral CT scans and thoracoscopy.

This is a prospective, multi-center, double-blind, statistically powered clinical trial that will enroll patients scheduled to undergo a procedure for removal of fluid from a pleural effusion (i.e. thoracentesis, thoracoscopy, image guided thoracentesis, thoracotomy, chest tube placement, Pleurex® catheter insertion, etc.).

The primary objective of the study is to evaluate the ability of multiple biomarkers in serum and/or pleural fluid to estimate the risk of finding cancer in subjects presenting with an undiagnosed pleural effusion (i.e. unknown origin).

The secondary objective of the study is to compare the ability of multiple biomarkers in serum and/or pleural fluid combined with pleural fluid cytology and other laboratory results to the use of the multiple biomarkers alone to estimate the risk of finding cancer in subjects presenting with an undiagnosed pleural effusion.

The research objectives of the study are the evaluation of the utility of multiple biomarkers in serum and/or pleural fluid to predict the tissue of origin in subjects with cancer who presented with an undiagnosed pleural effusion and comparison of these results to pleural fluid cytology. Correlation of the biomarker levels in the serum and pleural fluid will be evaluated as well.

ELIGIBILITY:
Inclusion Criteria:

TRAINING SET INCLUSION CRITERIA

* Subjects able to understand and sign Informed Consent;
* Males or females >18 years of age;
* Have a pleural effusion of known or unknown origin;
* Scheduled for a diagnostic and/or therapeutic procedure to remove pleural fluid.

VALIDATION SET INCLUSION CRITERIA

* Subjects able to understand and sign Informed Consent;
* Males or females >18 years of age;
* Have a pleural effusion of unknown origin;
* Scheduled for a diagnostic procedure to remove pleural fluid.

Exclusion Criteria:

TRAINING SET EXCLUSION CRITERIA

* For Subjects currently receiving chemotherapy and/or radiation therapy- Subjects who have received chemotherapy and/or radiation therapy must have completed these modalities one month before entering the study.
* Females known to be pregnant;
* Already entered into the study;
* Unable or unwilling to provide informed consent or is there a high risk that the subject may not comply with the protocol requirements

VALIDATION SET EXCLUSION CRITERIA

* For Subjects currently receiving chemotherapy and/or radiation therapy- Subjects who have received chemotherapy and/or radiation therapy must have completed these modalities one month before entering the study.
* Females known to be pregnant;
* Already entered into the study;
* Unable or unwilling to provide informed consent or is there a high risk that the subject may not comply with the protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: N/A - study was closed
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2006-03; Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Allard, PhD, Study Director — Fujirebio Diagnostics, Inc.
Locations (1):
- Fujirebio Diagnostics, Inc, Malvern, Pennsylvania, United States